CLINICAL TRIAL: NCT04100213
Title: Real-Time Assessment of Stress and Stress Response
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants were willing to enroll.
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Stephan T. Egger, Senior Psychiatrists, Psychiatric University Hospital, Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: mHealth TSST-G
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Psychiatric Disorder; Stress Reaction; Stress, Psychological; Stress, Physiological
Keywords: Stress, Stress Reaction, Trier Social Stress Test, Digital Phenotyping
MeSH Terms: conditions — Mental Disorders; Fractures, Stress; Stress, Psychological | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TSST (Experimental)
  Interventions: Behavioral: Trier Social Stress Test

INTERVENTIONS:
Behavioral: Trier Social Stress Test — The TSST-G is a psychological paradigm which combines high levels of social-evaluative threat and uncontrollability in a group setting. The TSST-G will proceed in groups of three to five participants (from the same diagnostic group). The TSST-G consists of three phases: a briefing; the psychological test itself, followed by a debriefing phase. Each phase will last 40, 20 and 60 minutes, respectively. The briefing and debriefing of the TSST-G will be conducted by experienced psychotherapists. The TSST-G itself will be conducted by personal unknown to the participants.
  Other Names: TSST

SUMMARY:
Stress is a complex natural phenomenon, frequently related to a physiological response, including heart rate, heart rate variability, respiratory rate, skin conductance and temperature. The subjective experience varies greatly; broadly, it may be conceived as a freeze, flight, fight, fright or faint response. Many studies have demonstrated the negative influence of psychological stress on health and well-being. Through the digital phenotyping of physiological and psychological stress reactions, in a controlled laboratory setting (Trier Social Stress Test- TSST) and real-life situations, in a population of healthy participants and patients with a major psychiatric disorder, we expect to find reliable and valid digital biomarkers. The results of this study will, therefore, not only contribute to a better understanding of stress and stress response but also have the potential to improve diagnostic and treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Participants are competent to give informed consent.
* Participants are right handed
* German language proficiency as a native speaker or level B1
* Diagnosis of a cluster C personality disorder according to ICD-10; or
* Diagnosis of depressive disorder according to ICD-10; or
* Diagnosis of schizophrenia or schizoaffective disorder according to ICD-10; or
* Without a current psychiatric disorder.

Exclusion Criteria:

* Low Intelligence as confirmed by failure to complete regular compulsory education.
* Pregnancy or over two weeks delay in the menstrual cycle.
* Previous participation in a psychological trial involving psychosocial stress assessment.
* Current neurological disorder.
* Current cardiovascular disorder.
* Current respiratory disorder.
* Current substance use or withdrawal.
* Any change in medication in the previous week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Cortisol | Change from 40 and 20 min. before the intervention. 0, 10, 20 30, 40, 60 and 80 min. after the intervention
  Saliva Cortisol Concentration
Subjective Stress | Change from 40 and 20 min. before the intervention. 0, 10, 20 30, 40, 60 and 80 min. after the intervention
  Stress Questionnaire

SECONDARY OUTCOMES:
Psychopathological Assessement | 1 day
  Symptom Questionnaire
Psychiatric Diagnosis | 1 day
  Structured psychiatric Interview

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egger ST, Knorr M, Bobes J, Bernstein A, Seifritz E, Vetter S. Real-Time Assessment of Stress and Stress Response Using Digital Phenotyping: A Study Protocol. Front Digit Health. 2020 Oct 15;2:544418. doi: 10.3389/fdgth.2020.544418. eCollection 2020. PMID 34713030